CLINICAL TRIAL: NCT04184141
Title: The Effect of Hydroxyzine and Alprazolam Premedication on Preoperative Anxiety and Patient Satisfaction
Brief Title: Preoperative Use of Alprazolam and Hydroxyzine in Anxiety
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Principal investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0195
Record Dates: First submitted 2019-11-30; First posted 2019-12-03 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Agitation on Recovery From Sedation
MeSH Terms: interventions — Hydroxyzine; Alprazolam

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- alprazolam (Experimental)
  Interventions: Drug: Alprazolam tablet
- hydroxyzine (Experimental)
  Interventions: Drug: Hydroxyzine Hydrochloride
- control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxyzine Hydrochloride — Hyroxyzine hydrochloride is given to the patient one hour before surgery.
  Arms: hydroxyzine
Drug: Alprazolam tablet — Alprozolam is given to the patient one hour before surgery.
  Arms: alprazolam
Drug: Placebo — Placebo candy
  Arms: control

SUMMARY:
Patients will be divided into three groups. Group H patients will be given 100 mg Hydroxyzine orally 1 hour before surgery while group A patients will receive 0.5 mg Alprazolam orally. group P will be placebo group. Amsterdam Preoperative Anxiety and Knowledge Scale (APAIS) anxiety scores will be evaluated and recorded 1 hour before surgery. APAIS score will be evaluated again in the the operation room before surgery started. After base measurements of patients are recorded with standard monitoring, spinal block will be performed with 15 mg Heavy Bupivacaine from the L2-L3 or L3-L4 levels of spinal cord in sting position. When T10 level sensory block and Bromage 0-1 neuromusculer block will be occured , surgery will be started. Heart rate, non-invasive arterial blood pressure and the degree of peripheral O2 saturation will be measured at 5 minutes interval throughout the operation. IOWA anesthesia satisfaction scale will also performed to the patients the day after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* sacrococcygeal dermoid cyst patients
* Saceptance of spinal anaesthesia
* between 18-60 years old patients
* ASA I-II

Exclusion Criteria:

* drug allergy
* BMI>35kg/m2
* psychiatric disorders
* serious renal and hepatic damage
* coagulation disorders
* serious cardiac and respiratory disorderders
* rejection of spinal anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
preopartive anxiety | 1 hour later orally admition of drugs
  Amsterdam Preoperative Anxiety and Information Scale (APAİS) (between 0-30)

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours after surgery
  IOWA pation satisfaction scale (between 9-54)

IPD SHARING:
Plan to Share IPD: No